CLINICAL TRIAL: NCT00415090
Title: Substitution by Nevirapine in HIV-1 Infected Patients on Triple Treatment of Reverse Transcriptase Nucleoside/Nucleotide Inhibitors
Brief Title: Study to Evaluate the Replacement of Reverse Transcriptase Nucleoside/Nucleotide Inhibitors by Nevirapine in Patients on Triple Treatment With Analogues Only
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Calella (Other)
Responsible Party: Hospital San Jaime de Calella, Hospital San Jaime de Calella
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIMUNE
Record Dates: First submitted 2006-12-19; First posted 2006-12-22 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections
Keywords: Nevirapine; Antiretroviral treatment; Triple nucleoside therapy; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Follow with same ARV treatment
- 2 (Experimental): Switch one of ARV drugs to Nevirapine
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Nevirapine — Switch one of ARV drugs to Nevirapine
  Other Names: Switch one of ARV drugs to Nevirapine
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the proportion of patients with viral load of HIV-1 < 50 copies after 48 weeks of follow-up after randomization to change or not to nevirapine.

DETAILED DESCRIPTION:
RTNI (reverse transcriptase nucleoside inhibitors) are a regular part of most antiretroviral combinations. The presence of a smaller or greater degree of cross resistance among all RTNI is increasingly better described and acknowledged, whereby the number of salvage regimens that may be built following the appearance of this resistance to these drugs is by no means unlimited.

This proactive treatment change in patients on RTNI-based regimens while the viral load is still suppressed would avoid the selective replication period under antiviral pressure following the failure of the regimen in which resistance-associated mutations accumulate. This therapeutic approach has demonstrated its effectiveness in clinical practice, albeit not in this scenario.

If we wait until the viral load is detectable there is sufficient evidence that resistance to RTNI will appear and that this resistance will compromise future salvage options.

To intensify with this proactive approach these combinations based on N/NNRTI (nucleotide analog), the NNRTI are an optimal alternative.There is vast experience with NVP in simplification/maintenance trials. In direct comparative simplification studies in patients with virological response, the response rates with NVP or EFV have shown no differences. With a relative risk (RR) of virological failure of 0.54 with regard to the continuation of PI (protease inhibitors), NVP is one of the best simplification treatment options in HIV-1-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients on triple treatment with 3 nucleoside analogues or transcriptase nucleotide inhibitors in virological suppression.
* Age >= 18 years.
* Confirmed diagnosis of HIV-1 infection.
* Viral load < 50 copies/ml over the previous six months, including at least two consecutive determinations.
* Value of ALT transaminase £ 2.5 times the normal value of the laboratory of each centre.
* Acceptance and signature of the informed consent form.

Exclusion Criteria:

* Pregnant women or those who intend to become pregnant in the study period.
* Having had an active infection in the previous month.
* Previous exposure to any reverse transcriptase non-nucleoside inhibitor (nevirapine, efavirenz or delavirdine).
* Simultaneous treatment with methadone.
* Patients with serious hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma viral load below 50 copies/mL . | after 48 weeks of follow-up

SECONDARY OUTCOMES:
Time to the appearance of viral load >50 copies/mL in both branches (two consecutive determinations with 4-week separation between both). | During the 48 weeks of follow-up.
Evolution of the CD4 lymphocyte count at 48 weeks. | during 48 weeks of follow-up
Pattern of mutations associated with resistance in patients presenting virological failure. | When there is a virological failure
Incidence of adverse clinical effects and laboratory alterations, giving rise or not to the withdrawal of the investigational treatment. | during the 48 weeks of follow-up
Incidence of AIDS-defining events (CDC C events, 1993). | during the 48 weeks of follow-up
Mortality by any cause. | during the 48 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Josep Mª Llibre, MD,PhD, Principal Investigator — Hospital Sant Jaume de Calella
Locations (17):
- Spain (17):
  - Hospital.Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Centre Penitenciari Brians, Barcelona, Barcelona
  - Hopsital de Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Sant Jaume de Calella, Barcelona, Barcelona
  - Centre Penitenciari Homes, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Centre Penitenciari Quatre Camins, Granollers, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital La Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital La Fe de Valencia, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza
  - Hospital de Tortosa, Tortosa